CLINICAL TRIAL: NCT02697461
Title: Multisegmented Foot Motion in Patients With Lateral Ankle Sprains and Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jay Hertel, PhD, ATC, Prinicipal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 18550
Record Dates: First submitted 2016-01-11; First posted 2016-03-03 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Injuries, Ankle; Sprain of Foot
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrinsic Foot Arm (Experimental): In arm 1, a randomized control trial will be used in the investigation of validity and reliability comparing multisegmented foot motion, clinical joint physiological and accessory motion, and morphologic foot measurements, and the effect of intrinsic foot strengthening on multisegmented foot function.
  Interventions: Other: Intrinsic Foot Strengthening
- Joint Mobilization Arm (Experimental): In arm 2, the investigation of group differences in clinical and laboratory measures of multisegmented foot motion and kinetics will use a case control design. A randomized controlled trial will be conducted in the study investigating joint mobilization, with the researcher performing the assessments and the provider performing the treatments blinded to group allocation
  Interventions: Other: Joint Mobilization

INTERVENTIONS:
Other: Intrinsic Foot Strengthening — Intrinsic foot strengthening is a commonly used intervention in clinic used to increase foot stability both in prevention of and in treatment of foot and ankle injury. Subjects allocated to the strengthening program will be educated in commonly used short foot exercises and "toe yoga" maneuvers that target the intrinsic muscles of the foot. No equipment will be required to perform the exercises.
  Arms: Intrinsic Foot Arm
Other: Joint Mobilization — Joint mobilization is a commonly used clinical intervention used to decrease pain and increase joint range of motion. In the treatment groups who present with joint hypomobility, a forefoot inversion maneuver with a dorsally applied pressure in the lateral midfoot and rearfoot stabilized will be applied at the barrier before the physiologic end range of motion. A second mobilization will be performed at the distal segment of the 1st Tarsometatarsal joint. These mobilizations will be performed by a board certified orthopaedic physical therapist with 14-yrs of practice experience. No equipment will be required to perform the joint mobilization.
  Arms: Joint Mobilization Arm

SUMMARY:
Lateral ankle sprains (LAS) and chronic ankle instability (CAI) are common musculoskeletal injuries that are a result of inversion injury during sport. The midfoot is frequently involved during inversion injury, is often overlooked during clinical examination, and maybe contributory to the development of CAI. The purpose of this study is to investigate multisegmented foot motion using a motion capture system, clinical joint physiological and accessory motion, and morphologic foot measurements in recreationally active men and women with and without a history of lateral ankle sprains and chronic ankle instability. Additionally, the effects of a joint mobilization intervention in patients with diminished multisegmented foot motion and intrinsic foot strengthening in healthy individuals will be investigated.

DETAILED DESCRIPTION:
Arm 1:The purpose of this arm of the study is to determine if foot muscle exercises change the function of the foot. Up to 25 people will be enrolled in this arm of the study at the University of Virginia.

Arm 2: The purpose of this arm of the study is to determine if joint mobilization applied to the middle part of the foot will effect function in people who are healthy, have a history of lateral ankle sprains (LAS), or have chronic ankle instability (CAI) and have joint stiffness. Up to 125 people will be enrolled in this arm of the study at the University of Virginia. CAI is a condition where symptoms from an ankle sprain last longer than one year. These symptoms include a feeling of looseness, feelings that the participant may roll the ankle, or repeated ankle sprains. This study may help clinicians prescribe simple exercises at home to help treat CAI. The participants are being asked to be in this study, because they are physically active (participate in some form of physical activity for at least 20 minutes per day, three days per week) and are not currently seeking medical treatment/therapy for LAS/CAI. Joint mobilization is a commonly used clinical intervention used to decrease pain and increase joint range of motion. The home exercises employed for this study are commonly used clinically in the treatment of foot and ankle problems and include a foot and calf stretch and standing on one foot for 60 seconds. The participant will be asked to perform these exercises three times daily throughout the course of the day.

The investigators hypothesize that joint mobilization will improve patient oriented outcomes and measures of joint mobility and excursion in individuals with impaired foot mobility immediately post intervention and at 1-week follow-up, but not at 4 weeks; and intrinsic foot strengthening will result in differences in morphologic measures and intrinsic muscle cross-section in healthy individuals following a 4 week home exercise program.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants

* Aged 18-50
* All subjects will be physically active: Participating in some form of physical activity for at least 20 min per day, three times per week.
* All subjects will have no history of ankle injury.

LAS participants

* Aged 18-50
* All subjects with a history of ankle sprains, no lingering symptoms or disability, not actively receiving treatment for their ankle sprain
* All subjects will be physically active: Participating in some form of physical activity for at least 20 min per day, three times per week.

CAI participants

* Aged 18-50
* CAI with a history of recurrent ankle sprains, with the first sprain occurring longer than 12 months ago. They will have lingering symptoms, and disability, but not actively receiving treatment for their CAI
* All subjects will be physically active: Participating in some form of physical activity for at least 20 min per day, three times per week.

Exclusion Criteria:

* Neurological or vestibular disorders affecting balance
* Currently seeking medical care for LAS/CAI
* History of prior ankle surgery
* History of ankle or foot fracture
* Diabetes mellitus
* Current self-reported disability due to lower extremity pathology that may adversely affect neuromuscular function
* Lumbosacral radiculopathy
* Soft tissue disorders including Marfan's syndrome and Ehlers-Dandros syndrome
* Absolute contraindications to manual therapy
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05-09 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes in midfoot frontal plane range of motion during stance phase of gait. | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Segmental motion will be assessed using motion capture and measured in degrees.
Changes in ultrasound thickness measures of the abductor hallucis | Arm 1: Baseline, 4 wks.
  Muscle thickness measures will be measured in cm.
Foot and Ankle Ability Measure (FAAM) | Arm 1: Baseline, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Patient Report Outcome of Foot and Ankle Function
Changes in ultrasound thickness measures of the flexor digitorum brevis | Arm 1: Baseline, 4 wks.
  Muscle thickness measures will be measured in cm.
Changes in thickness measures of the flexor hallucis brevis | Arm 1: Baseline, 4 wks.
  Muscle thickness measures will be measured in cm.

SECONDARY OUTCOMES:
Changes in Foot morphological measurements across loading conditions | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Measurement of foot length, truncated foot length, foot width, and arch height in cm.
Changes in Clinical Measures of forefoot frontal plane range of motion | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Measured with an inclinometer in degrees.
Changes in Clinical Measures of range of motion of first ray flexion/extension | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Measured with a goniometer in degrees.
Changes in Clinical Measures of joint laxity of the forefoot | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed manually using a 7 point categorical scale from 0=ankylosed to 6=joint instability
Changes in Clinical Measures of joint laxity of the first ray | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed manually using a 7 point categorical scale from 0=ankylosed to 6=joint instability
Changes in Clinical Measures of toe flexor strength | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed using a handheld dynamometer in N
Changes in Clinical Measures of ankle inversion strength | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed using a handheld dynamometer in N
Changes in Clinical Measures of ankle eversion strength | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed using a handheld dynamometer in N
Changes in Clinical Measures of ankle dorsiflexion strength | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed using a handheld dynamometer in N
Changes in Clinical Measures of ankle plantarflexion strength | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Assessed using a handheld dynamometer in N
Star excursion balance test | Arm 1: Baseline, 1wk, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Clinical test of single limb reach/balance in the anterior, posterior lateral, and posterior medial directions in cm.
12-Item Short Form Survey from the RAND Medical Outcomes Study (VR-12) | Arm 1: Baseline, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Patient Report Outcome of Function
Visual Analogue Scale (VAS) | Arm 1: Baseline, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Patient Report Outcome of Pain
Godin leisure questionnaire | Arm 1: Baseline, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Patient Report Outcome of Physical Activity
11-item Tampa Scale of Kinesiophobia (TSK-11) | Arm 1: Baseline, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Patient Report Outcome of Kinesiophobia
Global Rate of Change (GROC) | Arm 1: Baseline, 5 wks. Arm 2: Baseline, 1wk, 2wks
  Patient Report Outcome of Change in Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hertel, PhD, ATC, Principal Investigator — University of Virginia
Locations (1):
- Exercise and Sports Injury Laboratory, University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Background] Feger MA, Herb CC, Fraser JJ, Glaviano N, Hertel J. Supervised rehabilitation versus home exercise in the treatment of acute ankle sprains: a systematic review. Clin Sports Med. 2015 Apr;34(2):329-46. doi: 10.1016/j.csm.2014.12.001. Epub 2015 Feb 14. PMID 25818717
- [Background] Delahunt E, Coughlan GF, Caulfield B, Nightingale EJ, Lin CW, Hiller CE. Inclusion criteria when investigating insufficiencies in chronic ankle instability. Med Sci Sports Exerc. 2010 Nov;42(11):2106-21. doi: 10.1249/MSS.0b013e3181de7a8a. PMID 20351590
- [Background] Gerber JP, Williams GN, Scoville CR, Arciero RA, Taylor DC. Persistent disability associated with ankle sprains: a prospective examination of an athletic population. Foot Ankle Int. 1998 Oct;19(10):653-60. doi: 10.1177/107110079801901002. PMID 9801078
- [Background] Braun BL. Effects of ankle sprain in a general clinic population 6 to 18 months after medical evaluation. Arch Fam Med. 1999 Mar-Apr;8(2):143-8. doi: 10.1001/archfami.8.2.143. PMID 10101985
- [Background] Konradsen L, Bech L, Ehrenbjerg M, Nickelsen T. Seven years follow-up after ankle inversion trauma. Scand J Med Sci Sports. 2002 Jun;12(3):129-35. doi: 10.1034/j.1600-0838.2002.02104.x. PMID 12135444
- [Background] Tanen L, Docherty CL, Van Der Pol B, Simon J, Schrader J. Prevalence of chronic ankle instability in high school and division I athletes. Foot Ankle Spec. 2014 Feb;7(1):37-44. doi: 10.1177/1938640013509670. Epub 2013 Nov 27. PMID 24287210
- [Background] Mok KM, Fong DT, Krosshaug T, Engebretsen L, Hung AS, Yung PS, Chan KM. Kinematics analysis of ankle inversion ligamentous sprain injuries in sports: 2 cases during the 2008 Beijing Olympics. Am J Sports Med. 2011 Jul;39(7):1548-52. doi: 10.1177/0363546511399384. Epub 2011 Apr 1. No abstract available. PMID 21460069
- [Background] Kristianslund E, Bahr R, Krosshaug T. Kinematics and kinetics of an accidental lateral ankle sprain. J Biomech. 2011 Sep 23;44(14):2576-8. doi: 10.1016/j.jbiomech.2011.07.014. Epub 2011 Aug 6. PMID 21824618
- [Background] Willems T, Witvrouw E, Delbaere K, De Cock A, De Clercq D. Relationship between gait biomechanics and inversion sprains: a prospective study of risk factors. Gait Posture. 2005 Jun;21(4):379-87. doi: 10.1016/j.gaitpost.2004.04.002. PMID 15886127
- [Background] Fong DT, Ha SC, Mok KM, Chan CW, Chan KM. Kinematics analysis of ankle inversion ligamentous sprain injuries in sports: five cases from televised tennis competitions. Am J Sports Med. 2012 Nov;40(11):2627-32. doi: 10.1177/0363546512458259. Epub 2012 Sep 11. PMID 22967824
- [Background] Fong DT, Chan YY, Mok KM, Yung PS, Chan KM. Understanding acute ankle ligamentous sprain injury in sports. Sports Med Arthrosc Rehabil Ther Technol. 2009 Jul 30;1:14. doi: 10.1186/1758-2555-1-14. PMID 19640309
- [Background] Wei F, Fong DT, Chan KM, Haut RC. Estimation of ligament strains and joint moments in the ankle during a supination sprain injury. Comput Methods Biomech Biomed Engin. 2015;18(3):243-8. doi: 10.1080/10255842.2013.792809. Epub 2013 May 8. PMID 23654290
- [Background] Bonnel F, Toullec E, Mabit C, Tourne Y; Sofcot. Chronic ankle instability: biomechanics and pathomechanics of ligaments injury and associated lesions. Orthop Traumatol Surg Res. 2010 Jun;96(4):424-32. doi: 10.1016/j.otsr.2010.04.003. Epub 2010 May 20. PMID 20493797
- [Background] Blakeslee TJ, Morris JL. Cuboid syndrome and the significance of midtarsal joint stability. J Am Podiatr Med Assoc. 1987 Dec;77(12):638-42. doi: 10.7547/87507315-77-12-638. No abstract available. PMID 3430355
- [Background] Fagel VL, Ocon E, Cantarella JC, Feldman F. Case report 183: dislocation of the cuboid bone without fracture. Skeletal Radiol. 1982 Jan;7(4):287-8. doi: 10.1007/BF00361989. No abstract available. PMID 7071629
- [Background] Littlejohn SG, Line LL, Yerger LB Jr. Complete cuboid dislocation. Orthopedics. 1996 Feb;19(2):175-6. doi: 10.3928/0147-7447-19960201-15. No abstract available. PMID 8834294
- [Background] Kollmannsberger A, De Boer P. Isolated calcaneo-cuboid dislocation: brief report. J Bone Joint Surg Br. 1989 Mar;71(2):323. doi: 10.1302/0301-620X.71B2.2925758. No abstract available.
- [Background] McDonough MW, Ganley JV. Dislocation of the cuboid. J Am Podiatry Assoc. 1973 Jul;63(7):317-8. doi: 10.7547/87507315-63-7-317. No abstract available. PMID 4146011
- [Background] Jacobsen FS. Dislocation of the cuboid. Orthopedics. 1990 Dec;13(12):1387-9. doi: 10.3928/0147-7447-19901201-12. No abstract available. PMID 2274483
- [Background] Gough DT, Broderick DF, Januzik SJ, Cusack TJ. Dislocation of the cuboid bone without fracture. Ann Emerg Med. 1988 Oct;17(10):1095-7. doi: 10.1016/s0196-0644(88)80453-0. PMID 3178001
- [Background] Drummond DS, Hastings DE. Total dislocation of the cuboid bone. Report of a case. J Bone Joint Surg Br. 1969 Nov;51(4):716-8. No abstract available. PMID 4984469
- [Background] Sondergaard L, Konradsen L, Holmer P, Jorgensen LN, Nielsen PT. Acute midtarsal sprains: frequency and course of recovery. Foot Ankle Int. 1996 Apr;17(4):195-9. doi: 10.1177/107110079601700402. PMID 8696494
- [Background] Martin RL, Davenport TE, Paulseth S, Wukich DK, Godges JJ; Orthopaedic Section American Physical Therapy Association. Ankle stability and movement coordination impairments: ankle ligament sprains. J Orthop Sports Phys Ther. 2013 Sep;43(9):A1-40. doi: 10.2519/jospt.2013.0305. No abstract available. PMID 24313720